CLINICAL TRIAL: NCT06548360
Title: A Phase 3, Randomized, Double-Blind, Safety, and Efficacy Study of Ruxolitinib Cream in Pediatric Participants With Nonsegmental Vitiligo
Brief Title: A Study to Evaluate the Safety and Efficacy of Ruxolitinib Cream in Pediatric Participants With Nonsegmental Vitiligo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB18424-312
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: NonSegmental Vitiligo
Keywords: NonSegmental Vitiligo; pediatric

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib 1.5 % Cream (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected area as defined in the protocol.
  Interventions: Drug: Ruxolitinib Cream
- Vehicle Cream (Placebo Comparator): Participants received vehicle cream, applied topically to the affected area as defined by the protocol.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.
  Other Names: INCB018424 Phosphate Cream
  Arms: Ruxolitinib 1.5 % Cream
Drug: Vehicle Cream — Matching vehicle cream applied topically to the affected area as a thin film twice daily.
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study is to to evaluate the safety and efficacy of ruxolitinib cream in pediatric participants with nonsegmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nonsegmental vitiligo with depigmented area including ≥ 0.5% BSA on the face, ≥ 0.5 F-VASI, ≥ 3% BSA on nonfacial areas, ≥ 3 T-VASI.
* Total body vitiligo area does not exceed 10% BSA.
* Pigmented hair within some of the areas of vitiligo on the face.
* Must agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit.
* For sexually active participants (except participants who are prepubescent) willingness to avoid pregnancy or fathering a child from screening through 30 days after the last application of study cream.

Exclusion Criteria:

* Diagnosis of other forms of vitiligo (eg, segmental).
* Other differential diagnosis of vitiligo or other skin depigmentation disorders (eg, piebaldism, pityriasis alba, leprosy, postinflammatory hypopigmentation, progressive macule hypomelanosis, nevus anemicus, chemical leukoderma, and tinea versicolor).
* Any other skin disease that, in the opinion of the investigator, would interfere with the study drug application or study assessments.
* Prior or current use of depigmentation treatments (eg, monobenzone).
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including application of study cream and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Use of protocol-defined treatments within the indicated washout period before baseline.
* Current or previous use of JAK inhibitors, systemic or topical.
* Protocol-defined clinically significant abnormal laboratory values at screening.
* BMI-for-age < 5th percentile or ≥ 85th percentile according to the CDC BMI Percentile Calculator for Child and Teen.
* Pregnant or lactating participants or those considering pregnancy during the period of their study participation.
* In the opinion of the investigator, unable or unlikely to comply with the application schedule and study evaluations.
* Living with anyone participating in any current Incyte-sponsored ruxolitinib cream study.
* Employees of the sponsor or investigator or are otherwise dependents of them.
* Known allergy or reaction to any component of the study cream formulation.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving a ≥ 75% Improvement From Baseline in the Facial Vitiligo Area Scoring Index (F-VASI75) | Week 24
  ≥75% improvement in facial Vitiligo Area Scoring Index.

SECONDARY OUTCOMES:
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI50) | Week 24
  ≥50% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI90) | Week 24
  ≥90% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving a ≥ 50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 24
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Percentage change from baseline in F-BSA | Week 24
  Facial body surface area (F-BSA) takes into account the facial depigmented areas as a percentage of the total body area.
Number of Treatment Emergent Adverse Events (TEAEs) | Up to Week 52 and 30 days
  TEAE defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI50) | Week 52
  ≥50% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI75) | Week 52
  ≥75% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI90) | Week 52
  ≥90% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 52
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI25) | Week 24 and Week 52
  ≥25% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI75) | Week 24 and Week 52
  ≥75% improvement in total body Vitiligo Area Scoring Index
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI90) | Week 24 and Week 52
  ≥90% improvement in total body Vitiligo Area Scoring Index
Pharmacokinetic (PK) of Ruxolitinib: Trough concentrations | Weeks 6, 24, 30 and 52
  Trough is defined as the concentration reached by a drug immediately before the next dose is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (99):
- United States (80):
  - University of Alabama At Birmingham-School of Medicine, Birmingham, Alabama
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Omni Dermatology, Phoenix, Arizona
  - Affiliated Dermatology, Scottsdale, Arizona
  - Banner - University Medicine Multispecialty Services Clinic, Tucson, Arizona
  - Premier Dermatology Clinical Trials Institute At Northwest Arkansas, Fayetteville, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Axon Clinical Research, Inglewood, California
  - University of California Irvine, Irvine, California
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - La Universal Research Center, Inc, Los Angeles, California
  - Stanford School of Medicine, Palo Alto, California
  - Empire Clinical Research, Pomona, California
  - Norcal Clinical Research, Rocklin, California
  - Peninsula Research Associates Pra, Rolling Hills Estates, California
  - Integrative Skin Science and Research, Sacramento, California
  - Rady Children'S Hospital-San Diego, San Diego, California
  - Children'S Hospital Colorado, Aurora, Colorado
  - Paradigm Clinical Research Centers, Inc., Wheat Ridge, Colorado
  - Skin Care Research, Llc, Boca Raton, Florida
  - Encore Medical Research, Llc Boynton Beach, Boynton Beach, Florida
  - Skin Care Research, Llc, Hollywood, Florida
  - Solutions Through Advanced Research, Inc, Jacksonville, Florida
  - Pediatric Skin Research Llc, Miami, Florida
  - Nicklaus Children'S Hospital, Miami, Florida
  - Dh Tamarac Research Center Etna Medical Center Emc, Tamarac, Florida
  - Usf Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Cleaver Medical Group, Cumming, Georgia
  - Advanced Medical Research Pc, Sandy Springs, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Illinois Dermatology Institute the Chicago Loop, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Forefront Dermatology, Libertyville, Illinois
  - Advanced Dermatology Lincolnshire, Lincolnshire, Illinois
  - Northshore University Healthsystem, Skokie, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Wellskin Dermatology & Aesthetics, Bowling Green, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Dermatology Associates Pc, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Michigan Center For Research Company, Clarkston, Michigan
  - Mi Skin Center, Pllc, Northville, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Boeson Research, Missoula, Montana
  - Skin Specialists Pc the Advanced Skin Research Center, Omaha, Nebraska
  - The University of New Mexico Unm Health Sciences Center Hsc, Albuquerque, New Mexico
  - Suny Downstate Medical Center, Brooklyn, New York
  - The Dermatology Specialists Greenwich, New York, New York
  - Equity Medical, Llc, New York, New York
  - Mount Sinai Doctors, New York, New York
  - Sadick Dermatology Sadick Research Group, New York, New York
  - Skin Search of Rochester, Rochester, New York
  - Vitality Clinical Research Llc, Woodbury, New York
  - Red River Research Partners, Fargo, North Dakota
  - Dermatologists of Southwestern Ohio, Llc, Bexley, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Columbia Dermatology, Columbia, South Carolina
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Dell Children'S Medical Group, Austin, Texas
  - The University of Texas Health Science Center At Houston, Bellaire, Texas
  - Dfw Clinical Trials, Carrollton, Texas
  - 3A Research Llc West Location, El Paso, Texas
  - Reveal Research Institute, Frisco, Texas
  - Acrc Trials, Grapevine, Texas
  - Us Dermatology Partners Longview, Longview, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Stryde Research, Southlake, Texas
  - University of Utah Midvalley Dermatology, Murray, Utah
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Virginia Clinical Research, Inc Vcr Pariser Dermatology Specialists, Ltd Norfolk Location, Norfolk, Virginia
  - Frontier Dermatology, Mill Creek, Washington
  - Seattle Children'S Hospital, Seattle, Washington
  - Dermatology Specialists of Spokane, Spokane, Washington
  - University of Wisconsin School of Medicine, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (19):
  - Kirk Barber Research, Calgary, Alberta
  - Dermatology Research Institute, Calgary, Alberta
  - Alberta Health Services (Ahs) - Alberta Children'S Hospital (Ach), Calgary, Alberta
  - Laser Rejuvenation Clinics Edmonton D.T. Inc, Edmonton, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - Coal Harbour Rejuvenation Dermatology, Inc., Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Maritime Dermatology, Halifax, Nova Scotia
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - Dar Clinical Research Inc, Ottawa, Ontario
  - University of Toronto - the Hospital For Sick Children (Sickkids), Toronto, Ontario
  - Dermatelier on Avenue, Toronto, Ontario
  - Cosmetic Dermatology on Bloor, Toronto, Ontario
  - Centre de Recherche St-Louis, Montreal, Quebec
  - Universite de Montreal - Centre Hospitalier Universitaire (Chu) Sainte-Justine - Centre de Recherche, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec - Centre Hospitalier de L'Universite Laval (Chul), Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
  - Skincare Studio Dermatology Centre, St. John's

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Safety and Efficacy of Ruxolitinib Cream in Pediatric Participants With Nonsegmental Vitiligo — https://incyteclinicaltrials.com/studies/incb18424-312